CLINICAL TRIAL: NCT06872593
Title: Validating a Novel Driving Simulation-based MWT Against the Standard MWT in an OSA-cohort Challenged by CPAP-withdrawal - a Monocentric, Controlled, Randomized, Crossover Trial
Brief Title: Validating a Novel Driving Simulation-based MWT Against the Standard MWT in an OSA-cohort Challenged by CPAP-withdrawal
Acronym: DS-MWT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stefan Lakämper (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor-Investigator, Stefan Lakämper, Dr. rer. nat. , Head Research & Research Development, Division of TRaffic Medicine, Institute for Forensic Medicine, University of Zurich, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DS-MWT2
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-03

CONDITIONS: Excessive Daytime Sleepiness; Obstructive Sleep Apnea (OSA); CPAP Treatment; Driving Simulator Performance; Driving Impaired; CPAP
Keywords: sleep; drowsy driving; sleepy driving; sleepiness behind the wheel; driving simulation; CPAP treatment; CPAP withdrawal; driving performance; sleep latency; maintenance of wakefulness test; MWT; microsleep; microsleep-like episodes; eye tracking; EEG-recording
MeSH Terms: conditions — Disorders of Excessive Somnolence; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: monocentric, controlled, randomized, crossover trial, with two groups and four arms, plus a two-armed crossover control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- OSA - W(first) + MD (Experimental): allocated OSA-participants will perform test sequence M -> D first after 7d CPAP-withdrawal, then after ≥7d CPAP.
  Interventions: Procedure: CPAP-withdrawal; Diagnostic Test: Test Sequence
- OSA - W(first) + DM (Experimental): allocated OSA-participants will perform test sequence D -> M first after 7d CPAP-withdrawal, then after ≥7d CPAP.
  Interventions: Procedure: CPAP-withdrawal; Diagnostic Test: Test Sequence
- OSA - C(first) + MD (Experimental): allocated OSA-participants will perform test sequence M -> D first after ≥7d CPAP, then after 7d CPAP-withdrawal.
  Interventions: Procedure: CPAP-withdrawal; Diagnostic Test: Test Sequence
- OSA - C(first) + DM (Experimental): allocated OSA-participants will perform test sequence D-> M first after ≥7d CPAP, then after 7d CPAP-withdrawal.
  Interventions: Procedure: CPAP-withdrawal; Diagnostic Test: Test Sequence
- Healthy control MD - DM (Other): healthy participants will perform test sequence M -> D first , then D -> M
  Interventions: Diagnostic Test: Test Sequence
- Healthy control DM - MD (Other): healthy participants will perform test sequence D -> M first , then M -> D.
  Interventions: Diagnostic Test: Test Sequence

INTERVENTIONS:
Procedure: CPAP-withdrawal — 7-day-long CPAP-withdrawal
  Arms: OSA - C(first) + DM; OSA - C(first) + MD; OSA - W(first) + DM; OSA - W(first) + MD
Diagnostic Test: Test Sequence — Test Sequence M or D as specified in arm description

SUMMARY:
In brief, the proposed study will evaluate a recently proposed naturalistic, driving simulation test to identify and measure sleepiness behind the wheel, one of the most underestimated causes of road accidents. The proposed test offers higher ecological validity and might complement somnological tests that are standard, but rarely performed. Thus, the test might provide traffic medicine and sonologists with an effective tool, that can also directly convey the risks of excessive daytime sleepiness to drivers and thus, in combination, effectively aid in traffic medicine's mandate to avoid preventable road fatalities.

Excessive daytime sleepiness (EDS) is a symptomatic condition resulting from too little or compromised sleep, caused by psycho-social stress (shiftwork, lifestyle) or medical conditions (obstructive sleep apnoea (OSA), narcolepsy). Driving with untreated EDS might lead to sleepy/drowsy driving and microsleep, which is considered to be one of the highest-ranking causes of road accidents. Sleepiness and its dangers on the wheel might subjectively not be registered by the affected drivers. Also, subjective sleepiness might not correlate with somnological measurements that are also crucial for legally determining the fitness to drive (FTD).

There exists a variety of partially complementary tools to evaluate the extent of EDS. Mean sleep latency obtained in the maintenance of wakefulness test (MWT) is widely, but not uniformly, considered to be one of the most objective measures to evaluate EDS, especially in the context of driving performance. However, there is inconsistent or insufficient evidence for MWTs to reliably predict the FTD in general, potentially as its result might be strongly influenced by motivation. Moreover, patients might not relate low mean MWT-latencies to their own and other's risks in traffic.

A need for improved tools to measure EDS was formulated. It remains open, whether the MWT should be replaced or complemented by, for example, future road-side metabolomics-tests detecting sleepiness in traffic or whether the MWT should be adapted to better convey a.) the risks of EDS in traffic and b.) its meaning for the determination of the FTD.

With this need in mind the investigators proposed furnishing the maintenance of wakefulness test with improved ecological validity to provide an improved tool for the assessment of the effect of excessive daytime sleepiness on the fitness to drive: recently published results from an exploratory feasibility study suggested it to be well possible to transfer the MWT-paradigm to a driving simulator (DS) with high user acceptance. The published result's implication and relevance was well received: the new test, DS-MWT, might complement somnological MWTs in pneumology and neurology. I might provide a naturalistic and relatable tool to determine EDS in traffic medicine, who is institutionally responsible for determining the FTD. This is also desirable, because prohibitively high cost - in time, money and instrumentation - often prevent a standard MWT in standard care of sleep-related medical conditions. Potentially, the use of the DS-MWT might help reduce the number of preventable road fatalities by more often identifying sleepy individuals before they get behind the wheel.

However, for this goal to be achieve, it remains to be evaluated whether the latencies obtained in classical or simulation conditions are comparable and whether obtained latencies actually reflect other clinical parameters of EDS relating to underlying medical conditions, such as for example OSA. This represents a significant gap of evidence for both medical experts in pneumology and traffic medicine, but also for affected drivers. This gap will be filled by systematically comparing classical and simulation-based MWTs by means of their resulting latencies. In a within-study setup of 36 highly adherent OSA-patients, experiments will be related to a main medical comparator, a ≥7-day continuous positive airway pressure (CPAP)-withdrawal (W) and subsequent -resumption or continuation (C), respectively. There will be a control group of 18 healthy participants for comparison.

ELIGIBILITY:
Inclusion Criteria (OSA patients): adult drivers, diagnosed OSA, established CPAP-treatment regime, highly adherent and compliant within the last 6 months (>5h, >80% of days), at impaired eyesight with more than +/- 5 diopter or astigmatism, contact lenses are required (for eye tracking)

Inclusion criteria (healthy comparison croup): adult drivers, no declared psychiatric disorders, no declared sleep-related diagnosis, at impaired eyesight with more than +/- 5 diopter or astigmatism, contact lenses are required (for eye tracking)

Exclusion criteria (for both groups): sensibility to motion sickness (kinetosis, dizziness, etc. in 5 min screening drive), professional drivers (if working during the study period), inability to understand the study procedure for linguistic or cognitive reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
significant difference between mean MWT- and DS-MWT-latencies | MWT- and DS-MWT-latencies are measured in two consecutive days during CPAP-treatment and after 7 days CPAP-withdrawal (intervention) in randomized order.
  significant difference between mean latencies measured in classical maintenance of wakefulness test (MWT, M) and driving simulation-based maintenance of wakefulness test (DS-MWT, D) and DS-MWT-latencies.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lakämper, Dr. rer. nat., Principal Investigator — University of Zurich; Esther I Schwarz, PD, Dr. med., Principal Investigator — University of Zurich; Kristina Keller, Dr. med., Principal Investigator — University of Zurich
Locations (1):
- Division of Traffic Medicine, Institute of Forensic Medicine, University of Zurich, Zurich, ZRH, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in peer-reviewed journals. Anonymized raw data will be made available upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: starting after publication of study protcol and/or results
Access Criteria: upon request by mail

REFERENCES:
- [Background] Pisteljic M, Keller K, Lakamper S. Capturing sleep accidents in driving simulation as a promising tool to assess excessive daytime sleepiness with high ecological validity-a pilot study. Sleep. 2024 Aug 14;47(8):zsae110. doi: 10.1093/sleep/zsae110. No abstract available. PMID 38758109
- See also: Swiss National Clinical Trial Prortall (SNCTP) Registration of DS-MWT2 — https://www.humanforschung-schweiz.ch/de/studiensuche/studien-detail/66469/